CLINICAL TRIAL: NCT01870323
Title: The Social Media and Activity Research in Teens Trial
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13019
Record Dates: First submitted 2013-02-01; First posted 2013-06-06 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART Behavioral Group (Experimental): Intervention condition which has access to SMART Group Wall on Facebook and receives privately-delivered weekly behavioral modules. (SMART Facebook Group + video-based behavioral modules)
  Interventions: Behavioral: SMART Behavioral Group
- SMART Informational Group (Active Comparator): Comparison condition (i.e., attentional control) has access to SMART Group Wall on Facebook, and receives privately-delivered weekly text-based messages with generic content. (SMART Facebook Group + NO video-based behavioral modules)
  Interventions: Behavioral: SMART Informational Group

INTERVENTIONS:
Behavioral: SMART Behavioral Group — Test the efficacy of using social media to deliver a physical activity intervention based on social cognitive principles to increase lifestyle physical activity in low-active adolescents (i.e., access to regularly posted physical activity content on a study-specific, restricted access Facebook Group, as well as receipt of weekly video-based behavioral modules).
  Arms: SMART Behavioral Group
Behavioral: SMART Informational Group — Test the efficacy of using social media to deliver a physical activity intervention to increase lifestyle physical activity in low-active adolescents (i.e., access to regularly posted physical activity content on a study-specific, restricted access Facebook Group, but does not receive the weekly video-based behavioral modules).
  Arms: SMART Informational Group

SUMMARY:
In an effort to address the physical inactivity crisis among adolescents, the present study will examine the efficacy of using an already established Web-based social networking platform (i.e., Facebook) to deliver a physical activity intervention to adolescents.

DETAILED DESCRIPTION:
In an effort to address the physical inactivity crisis among adolescents, the present study will examine the efficacy of using an already established Web-based social networking platform (i.e., Facebook) to deliver a physical activity intervention to adolescents. The primary objectives of this trial are to 1) test the efficacy of a social media-delivered physical activity program for increasing lifestyle physical activity in adolescents, and 2) determine the effectiveness of a physical activity intervention based on social cognitive principles in comparison to a simple information-based physical activity condition. Additional objectives include an examination of how program participation may influence psychosocial health and how these changes affect physical activity patterns in youth.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 13-15 years of age
* Must not regularly meet nor exceed 60 minutes of daily physical activity
* Must have access to computer with Internet connection at home
* Must reside in Champaign County

Exclusion Criteria:

* Physical limitations that may prevent regular participation in physical activity or may inadvertently exacerbate any per-existing medical condition

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity | Baseline, Week 8, 4-Week Follow-Up (i.e., Week 12)
  Assessed objectively via accelerometry; subjectively via questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — Kinesiology & Community Health, UIUC
Locations (1):
- Exercise Psychology Laboratory, Urbana, Illinois, United States

REFERENCES:
- [Derived] Wojcicki TR, Grigsby-Toussaint D, Hillman CH, Huhman M, McAuley E. Promoting Physical Activity in Low-Active Adolescents via Facebook: A Pilot Randomized Controlled Trial to Test Feasibility. JMIR Res Protoc. 2014 Oct 30;3(4):e56. doi: 10.2196/resprot.3013. PMID 25357008